CLINICAL TRIAL: NCT02871154
Title: Extending the Time Period Between the Injection of Chorionic Gonadotropin and Oocyte Pick-up as a Solution to Low Rate of Mature Oocyte and Poor Results in Assisted Reproduction
Brief Title: Extending the hCG OPU Interval
Acronym: DelOPU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0041-16-POR
Record Dates: First submitted 2016-08-14; First posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Delay (Experimental): Delaying oocyte pick up beyond 39 hours post hCG
  Interventions: Other: Delaying oocyte pick up beyond 39 hours post hCG

INTERVENTIONS:
Other: Delaying oocyte pick up beyond 39 hours post hCG — Unlike the traditional less-than 39 hours interval from hCG injection to oocyte pick up, we will extend the interval up to 47 hours

SUMMARY:
Our and others experience suggest that in some cases delaying oocyte pick up (OPU) for more than 39 hours after hCG injection may be of benefit.

We plan to apply this to 20 women in whom less than 20% of oocytes were found suitable for intracytoplasmic sperm injection. The delay will be for up to an interval of 47 hours from hCG to OPU.

DETAILED DESCRIPTION:
In IVF one encounters some women in whom a low percentage of oocytes are found in the metaphase II stage upon their retrieval. Following some incidents, in our experience as well as others', where women injected hCG too early but oocytes were still retrieved with high proportion of maturity, we decided to delay OPU intentionally in women who had low percentage oocyte maturity in previous cycles.

ELIGIBILITY:
Inclusion Criteria: Previous 2 oocyte pick up cycles with 20% metaphase II oocytes in the cohort -

Exclusion Criteria:

No previous IVF history

-

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Conception | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Odeh-L'ya Katz, PhD, Study Director — Beruch Padeh Med Ctr Research Authority

IPD SHARING:
Plan to Share IPD: Yes
Study results